CLINICAL TRIAL: NCT03669406
Title: Feasibility Study - The Place of Surgical Management by Fatty Autograft in Patients With Healed Pelvic Eschar. Interest in Secondary Prevention.
Acronym: FATSCAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 35RC17_8999_FATSCAR; 2017-A03022-51 (Other: N° ID-RCB)
Record Dates: First submitted 2018-09-10; First posted 2018-09-13 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Eschar
Keywords: Healed pelvic eschar; Paraplegic patient; Fat autograft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autograft fat (Experimental): Paraplegic patients with healed pelvic eschar
  Interventions: Procedure: Autograft fat

INTERVENTIONS:
Procedure: Autograft fat — autograft fat

SUMMARY:
Autografting of fat cells is widely used in plastic surgery in breast reconstruction, burn scars, unsightly scars etc. It is known that the autografting of fat cells not only makes it possible to bring adipocytes, and thus to create a volume, but also promotes neo-angiogenesis by providing the growth factors which allows an improvement of the local cutaneous tissue.

Currently the investigators perform this action in their service on healed eschars, by analogy with burn scars that are also dystrophic, so as to improve cutaneous trophicity, and reduce the recurrence of eschars on these scars. However, the literature on the autografting of fat cells on eschars is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 65 years old;
* presenting a medullary, post-traumatic or congenital lesion, with consequent paraplegic sequelae;
* With a history of eschar:

  * Pelvic (ischiatic, trochanteric or sacral),
  * Healed for at least 6 months, after surgical treatment or directed healing (scarring is defined by the absence of local care, ie no nursing care);
* Affiliated to a social security ;
* Written informed consent.

Exclusion Criteria:

* Patient malnourished (albuminemia <40g / L);
* Non-weaning or weaned tobacco addiction for less than 3 weeks (compared to the date of surgery);
* Contraindication to MRI ;
* Protected person subject to legal protection (legal safeguards, guardianship, trusteeship), person deprived of liberty,
* Pregnant woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence of eschar | 12 months

SECONDARY OUTCOMES:
Time of occurrence of recurrence of eschar (censored criterion) | 12 months
POSAS scale score | 12 months
  Clinical evaluation
Vancouver score | 12 months
  Clinical evaluation
Improvement Vancouver score | 12 months
  Clinical evaluation
Number of recurrence of eschar | 12 months
  Clinical evaluation : non-recurrence
Evaluation of neovascularization | 12 months
  by Speckle laser doppler
Volumetric assessment | 12 months
  by contouring MRI
Analysis of pro-angiogenic genes expressed in the stromal vascular fraction of the injected fat | 12 months
  RNA PCR
Analysis of the stromal vascular fraction of the injected fat | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie AILLET, Principal Investigator — CHU Rennes; Cécile MEAL, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No